CLINICAL TRIAL: NCT06886841
Title: Stress Of Co-parents Related to A Traumatic Experience of Birth Across Switzerland
Brief Title: Parental Well-being After Childbirth in Switzerland
Acronym: SOCRATES
Status: Recruiting | Type: Observational
Sponsor: Laurent Gaucher (Other)
Responsible Party: Sponsor-Investigator, Laurent Gaucher, Professor, School of Health Sciences Geneva
Organization: School of Health Sciences Geneva (Other)
Other Study IDs: G700026130408; 220494 (Other Grant/Funding Number: Swiss National Science Foundation)
Record Dates: First submitted 2025-03-12; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Mental Health; Physical Health; Postpartum; Parents; Quality of Life; Quality of Care; Stress Disorder, Post Traumatic
Keywords: childbirth-related post-traumatic stress disorder; mental health; postpartum; parental wellbeing; physical health; sexual health; social support; quality of life; quality of care; postpartum depression; mothers; coparents
MeSH Terms: conditions — Psychological Well-Being; Stress Disorders, Post-Traumatic; Depression, Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Improving maternal and child health is a global priority, with increasing emphasis on ensuring women and their families not only survive but also thrive after childbirth. While high-income countries like Switzerland provide strong antenatal and intrapartum care, the quality of postnatal care often lags behind, despite the critical physical, mental, and social needs of the postpartum period. Studies indicate high rates of mental distress, physical pain, and sexual discomfort among mothers, alongside a lack of research on the well-being of co-parents.

The main question this cohort study aims to answer is: how do the health and well-being of mothers and co-parents evolve during the first year after childbirth? Participants will complete four online questionnaires: the first within the first few days after birth, followed by additional assessments at 2, 6, and 12 months postpartum.

This comprehensive approach seeks to inform policy and improve evidence-based postnatal care practices, benefiting approximately 80,000 families annually in Switzerland.

ELIGIBILITY:
Inclusion criteria:

* Women who give birth in a participating maternity unit or birth center during the study period.
* Partner of a participating women: the partner must be designated by the mother, live with her at the time of birth, and only one partner can be included per mother.
* Gestational age at birth: ≥22+0 weeks and/or birthweight ≥500 grams
* Age: Participants must be 14 years or older.
* Language Proficiency: Participants must have sufficient proficiency in one of Switzerland's main official languages (German, French, Italian) or English to ensure accurate communication and comprehension of study materials.

Exclusion Criteria:

* Refusal to participate
* Inability to provide informed consent

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All adult women who give birth to one or more live-born or stillborn children at ≥22 weeks and/or with a birthweight of ≥500 grams in a participating unit during the study period will be eligible, along with their cohabiting partners.
Sampling Method: Probability Sample
Enrollment: 4200 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Childbirth-related post-traumatic stress disorder | 2 months postpartum
  The prevalence of childbirth-related post-traumatic stress disorder in both parents will be assessed using the validated City Birth Trauma Scale (City BiTS). This self-reported questionnaire consists of 29 items, 20 of which measure the frequency of trauma symptoms, including intrusive thoughts, avoidance, negative mood, and hyperarousal, based on the criteria of the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5). Items are rated using a four-point Likert-type scale, ranging from 0 to 3. The total score varies from 0 to 60 points, with higher scores indicating a higher level of PTSD-symptoms.

SECONDARY OUTCOMES:
Postpartum depression and anxiety | At birth, and at 2, 6, and 12 months postpartum
  Postpartum depression and anxiety will be assessed in both parents, using the Edinburgh Postnatal Depression Scale (EPDS) at birth, and at 2, 6, and 12 months postpartum. This validated 10-item questionnaire screens for symptoms of depression and anxiety. Responses are rated on a four-point Likert scale, ranging from 0 to 3. The total score ranges from 0 to 30 points, with higher scores indicating a greater risk of depression.
Health-related quality of life | At birth, and at 2, 6, and 12 months postpartum
  Assessed in both parents with the EuroQoL 5-Dimension 5-Level scale (EQ-5D-5L), along with a visual analogue scale for self-rated health (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a visual analogue scale ranging from 0 to 100 where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
Physical recovery | At birth (Obstetric Quality of Recovery-10), and at 2, 6, and 12 months postpartum (pain and incontinence)
  Mothers' quality of recovery after childbirth, will be assessed using the Obstetric Quality of Recovery-10 (ObsQoR-10) tool. This validated, self-reported measure evaluates pain, physical symptoms, mobility, self-care, and baby care on an 11-point scale ranging from 0 (worst outcome) to 10 (best outcome). The total score ranges from 0 to 100, with higher scores indicating better recovery quality. Additional dimensions, in particular pain and incontinence, will also be evaluated in mothers.
Sexual health | 6 and 12 months postpartum
  Assessed at 6 and 12 months postpartum in mothers using the Female Sexual Function Index (FSFI-6), a validated questionnaire that can be used to screen for sexual dysfunction in women. It consists of 6 items covering 6 domains (desire, arousal, lubrication, orgasm, satisfaction, and pain). Each item of the FSFI-6 questionnaire is associated with a 5-point ordinal scale, in which 5 represents optimal function and 1 the poorest function. The scores for each domain are summed to provide a total score, with a higher score indicating better sexual function.
Hospitalisations | From one year before to one year after childbirth
  Collected through linkage with the "Medical Statistics of Hospitals" database, this outcome includes the frequency, reasons, and costs of hospitalisations from one year before to one year after childbirth. This data provides critical insights into severe health outcomes and rehospitalisations in mothers and infants.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Gaucher, RM, PhD, Principal Investigator — Geneva School of Health Sciences, HES-SO University of Applied Sciences and Arts Western Switzerland, Geneva, Switzerland.
Locations (2):
- Switzerland (2):
  - Haute Ecole de Santé Genève, Geneva
  - ZHAW Zurich University of Applied Sciences, Winterthur

IPD SHARING:
Plan to Share IPD: Yes
In compliance with the requirements of the Swiss National Science Foundation, anonymized study data will be made available to other researchers via Yareta, a certified and secure Swiss institutional research data repository. This ensures transparency, facilitates further research, and aligns with FAIR (Findable, Accessible, Interoperable, and Reusable) data principles. Access to the data on this platform is subject to authorization by a competent authority.
Supporting Information: Study Protocol, ICF
Time Frame: Undecided
Access Criteria: Researchers will have access to the IPD and supporting information. Data access via the YARETA platform is subject to authorization by a competent authority.
URL: https://yareta.unige.ch/